CLINICAL TRIAL: NCT07082660
Title: A Randomized Controlled Trial On Lumbal Disc Herniation Using Tecar Therapy: Effects On Pain And Functionality
Brief Title: Tecar Therapy in Lumbar Disc Herniation
Acronym: LDH-TECAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Şebnem Nur Alkan (Other)
Responsible Party: Sponsor-Investigator, Şebnem Nur Alkan, Assistant Professor of Physiotherapy, Atlas University, Atlas University
Organization: Atlas University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ETTBI-LDH-2023-01
Record Dates: First submitted 2025-07-15; First posted 2025-07-24 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Lumbal Disc Herniation; Capacitive and Resistive Electric Transfer Therapy; Exercise Training
Keywords: Lumbal disk herniation; Capasitive and resistive electric transfer therapy; exercise training

STUDY DESIGN:
Intervention Model Description: Participants were randomly assigned to two parallel groups receiving either TECAR + lumbar stabilization or lumbar stabilization only.
Who Masked: Participant
Masking Description: Participants were masked to their group assignments throughout the intervention period. Both groups received treatment in a similar clinical environment, and the application of TECAR therapy was performed using identical procedures and equipment setup to prevent participants from discerning their allocation. The physiotherapist administering the intervention was aware of group assignments, but outcome assessments were standardized to minimize bias.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TECAR Therapy Combined with Lumbal Stabilization Exercises (Experimental): Participants in this group will receive high-frequency capacitive-resistive diathermic current (TECAR) therapy (20 minutes per session, 3 sessions/week for 4 weeks) in addition to a lumbal stabilization exercise program (12 sessions total).
  Interventions: Device: High-Frequency Capacitive-Resistive Diathermic Current Therapy (TECAR)
- Lumbal Stabilization Exercises Only (Active Comparator): Participants in this group will receive only the lumbal stabilization exercise program, 3 sessions/week for 4 weeks (12 sessions total), with no TECAR therapy applied.
  Interventions: Behavioral: Lumbal Stabilization Exercise Program

INTERVENTIONS:
Device: High-Frequency Capacitive-Resistive Diathermic Current Therapy (TECAR) — 20 minutes per session, 3 times per week for 4 weeks
  Arms: TECAR Therapy Combined with Lumbal Stabilization Exercises
Behavioral: Lumbal Stabilization Exercise Program — 3 sessions per week for 4 weeks, each session includes core stabilization and lumbar control exercises (12 sessions total).
  Arms: Lumbal Stabilization Exercises Only

SUMMARY:
This randomized controlled trial investigates the effects of Tecar therapy on pain intensity and functional status in patients with lumbar disc herniation. The intervention group received Tecar therapy combined with conventional physiotherapy, while the control group received only conventional physiotherapy. Outcome measures include pain intensity, lumbar mobility, and functional disability. The study aims to determine whether Tecar therapy provides additional benefits compared to standard care in the early rehabilitation of individuals with lumbar disc herniation.

DETAILED DESCRIPTION:
Background Lumbar disc herniation (LDH) is a prevalent musculoskeletal condition that can significantly impair quality of life due to pain and functional limitations. Rehabilitation strategies often include lumbar stabilization exercises, and adjunct electrotherapies such as capacitive-resistive diathermy (TECAR) have gained interest for their potential therapeutic effects.

Purpose This randomized controlled trial aims to evaluate the effects of adding high-frequency capacitive-resistive diathermic current (TECAR) therapy to lumbar stabilization exercises, compared to lumbar stabilization exercises alone, on pain intensity, functional status, and lumbar range of motion in individuals with chronic LDH.

Methods

Thirty participants with chronic LDH (duration >6 months) and no neurological deficits will be randomly assigned to one of two intervention groups:

TECAR + Exercise Group (TEG, n=15): Participants will receive 12 sessions of TECAR therapy (20 minutes, 3 sessions per week) in combination with lumbar stabilization exercises over 4 weeks.

Exercise Group (EG, n=15): Participants will receive only lumbar stabilization exercises with the same frequency and duration.

Outcome measures will include:

Pain intensity (Visual Analog Scale - VAS)

Functional status (Oswestry Disability Index - ODI)

Lumbar range of motion (goniometry)

All evaluations will be performed pre- and post-intervention by a physiotherapist who is blinded to group allocation.

ELIGIBILITY:
Inclusion Criteria:

* aged 20-60 years
* diagnosed with low back pain
* pain localized between L1 and L5
* having low back pain lasting for more than 3 months [24].

Exclusion Criteria:

* having sensory disturbances
* muscle weakness, or reflex loss identified during motor, sensory, or reflex examinations
* history of prior lumbal spine surgery or vertebral fractures
* presence of electronic medical devices such as pacemakers or other implants contraindicated for electrical stimulation or high-frequency diathermy therapy
* patients officially registered as disabled or receiving social benefits due to low back pain, severe osteoporosis, osteomalacia, malignancy, infectious diseases, or systemic musculoskeletal or rheumatological disorders,
* pregnancy,
* cardiovascular conditions preventing exercise, or viscerogenic causes of low back pain

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-03-30 (Actual); Study Completion 2023-05-20 (Actual)

PRIMARY OUTCOMES:
Lumbar functionality | Baseline - 4 weeks
  The Oswestry Disability Index (ODI), validated Turkish version, will be used to assess disability related to low back pain. The scale consists of 10 items, each scored from 0 to 5, with a total maximum score of 50. The total score is converted into a percentage using the formula: (total obtained score / maximum possible score) × 100. Scores range from 0% to 100%, where higher scores indicate greater disability. Interpretation categories are as follows: 0%-20% indicates minimal disability; 21%-40% indicates moderate disability; 41%-60% indicates severe disability; 61%-80% indicates crippled; and 81%-100% indicates bed-bound status or possible symptom exaggeration.

SECONDARY OUTCOMES:
Pain intensity | Baseline - 4 weeks
  The Visual Analog Scale (VAS) will be used to assess pain intensity. It consists of a 10-centimeter horizontal line representing a continuum from 'no pain' (0) to 'worst imaginable pain' (10). Participants are asked to mark a point on the line that corresponds to the intensity of their pain. The distance in centimeters from the 'no pain' anchor to the participant's mark is measured and recorded as the VAS score. Scores range from 0 to 10, with higher scores indicating greater pain severity.

CONTACTS AND LOCATIONS:
Locations (1):
- Atlas University, Istanbul, Kagıthane, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) that underlie the results reported in the article (after deidentification) will be shared with other researchers upon reasonable request.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The IPD and supporting documents will be available beginning 6 months after publication of the primary results and will be accessible for a period of 3 years.